CLINICAL TRIAL: NCT05814627
Title: A Phase 3b/4 Randomized, Double-Blind, Double Dummy, Active Comparator-Controlled Study, Comparing the Efficacy and Safety of Upadacitinib Versus Adalimumab in Subjects With Moderate to Severe Rheumatoid Arthritis on a Stable Background of MTX and Who Had an Inadequate Response or Intolerance to a Single TNF Inhibitor (SELECT- SWITCH)
Brief Title: Study to Assess Change in Disease Activity and Adverse Events of Oral Upadacitinib Compared to Subcutaneous Adalimumab in Adult Participants With Moderate to Severe Rheumatoid Arthritis
Acronym: SELECT- SWITCH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-700; 2022-502578-18-00 (Other: EU CT)
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; Upadacitinib; Adalimumab; Methotrexate; MTX; TNF Inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upadacitinib+ Adalimumab matching Placebo (Experimental): Participants will receive upadacitinib once a day along with matching placebo for adalimumab at eow (every other week) in Period 1. Eligible participants will continue to receive same study treatment in Period 2 as assigned in Period 1.
  Interventions: Drug: Upadacitinib; Drug: Adalimumab Matching Placebo
- Adalimumab + Upadacitinib matching Placebo (Experimental): Participants will receive adalimumab at eow (every other week) along with matching placebo for upadacitinib once a day in Period 1. Eligible participants will continue to receive same study treatment in Period 2 as assigned in Period 1.
  Interventions: Drug: Adalimumab; Drug: Upadacitinib Matching Placebo

INTERVENTIONS:
Drug: Upadacitinib — Oral Tablets
  Other Names: RINVOQ
  Arms: Upadacitinib+ Adalimumab matching Placebo
Drug: Adalimumab — Subcutaneous Injection
  Other Names: Humira
  Arms: Adalimumab + Upadacitinib matching Placebo
Drug: Upadacitinib Matching Placebo — Oral Tablets
  Arms: Adalimumab + Upadacitinib matching Placebo
Drug: Adalimumab Matching Placebo — Subcutaneous Injection
  Arms: Upadacitinib+ Adalimumab matching Placebo

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease causing pain, stiffness, swelling and loss of joint function. This study will assess how safe and effective upadacitinib is in treating RA when compared to adalimumab in adult participants with inadequate response or intolerance to one TNF-inhibitor who are on a stable dose of methotrexate (MTX). Adverse events and change in disease activity will be assessed.

Upadacitinib is an approved drug for the treatment of RA. This study is double-blinded means that neither the participants nor the study doctors will know who will be given upadacitinib and who will be given adalimumab. Study doctors put the participants in 1 of the 2 groups, called treatment arms randomly, to receive either upadacitinib or adalimumab. There is 1 in 2 chance that participants will receive adalimumab. Each group consists of 2 periods. Approximately 480 participants diagnosed with RA will be enrolled in approximately 250 sites across the world.

Participants will receive the oral upadacitinib once daily and matching adalimumab placebo every other week, or the subcutaneous adalimumab every other week and matching upadacitinib placebo once daily during Period 1. Eligible participants will continue to receive same study treatment in Period 2 as assigned in Period 1 and will be followed for 30 days and 70 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis (RA) for >= 3 months based on the 2010 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) classification criteria for RA.
* Treated for >= 3 consecutive months prior to screening with 1 tumor necrosis factor inhibitor (TNFi) (only 1 of originator or biosimilar certolizumab pegol, etanercept, golimumab or infliximab) for RA, but continue to exhibit active RA, or had to discontinue due to intolerability or toxicity, irrespective of treatment duration. Up to 15% of participants who were intolerant to 1 TNFi will be allowed to enroll. Prior administration of different biosimilar versions for the same originator TNFi or switching between originator and biosimilar version of the same originator TNFi are acceptable. Cycling between biosimilars of different originator TNF inhibitors is not acceptable.
* On oral or parenteral methotrexate (MTX) therapy >= 3 consecutive months and on a stable prescription of 15 to 25 mg/week (or >= 10 mg/week in participants intolerant of MTX at doses >= 15 mg/week) for >= 4 weeks prior to the first dose of study drug. In addition, all participants should take a dietary supplement of folic acid or folinic acid throughout the study participation.

  * For a Chinese, Japanese, Korean, or Taiwanese participant, a stable dose of MTX >= 7.5 mg/week is acceptable.
  * Additional local requirements for MTX may apply.
* Meets both of the following disease activity criteria:

  * >= 6 swollen joint (based on 66 joint counts) and >= 6 tender joints (based on 68 joint counts) at screening and baseline;
  * High-sensitivity C-reactive protein (hsCRP) >= 3 mg/L (central lab, upper limit of normal [ULN] 2.87 mg/L) at screening.

Exclusion Criteria:

* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than Rheumatoid Arthritis (RA).
* Prior exposure to any janus kinase (JAK) inhibitor.
* Prior exposure to adalimumab (original or biosimilar) or to any approved or investigational TNF inhibitor other than infliximab, etanercept, certolizumab pegol and golimumab.
* Prior exposure to an approved or investigational non-TNFi biologic disease modifying anti-rheumatic drug (bDMARD) or targeted synthetic disease modifying antirheumatic drug (tsDMARD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Disease Activity Score 28 C-reactive Protein [DAS28-CRP]) <= 3.2 | Week 12
  The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. Low Disease Activity (LDA) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than or equal to 3.2.
Number of Participants with Adverse Events | From first dose of study drug until 70 days following last dose of study drug (up to approximately 58 weeks)
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.

SECONDARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology 50 % (ACR50) Response | Week 12
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  * 50% improvement in tender joint count (TJC68);
  * 50% improvement in swollen joint count (SJC66); and
  * 50% improvement in at least 3 of the 5 following parameters:
    * Physician's Global Assessment of Disease Activity measured on a Numerical Rating Scale of 0 to 10 (NRS)
    * Patient's Global Assessment of Disease Activity (NRS)
    * Patient's Assessment of Pain (NRS)
    * Health Assessment Questionnaire - Disability Index (HAQ-DI)
    * High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants Achieving Disease Activity Score 28 C-reactive Protein [DAS28-CRP]) < 2.6 | Week 12
  The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. Clinical remission (CR) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than 2.6.
Change from Baseline in Disease Activity Score 28 C-reactive Protein [DAS28-CRP]) | Week 12
  The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (NRS), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity.
Change from Baseline in Participants Assessment of Pain | Week 12
  Participants indicated their level of pain over the last 7 days using the Patient's Global Assessment Pain NRS. The range is 0 to 10 with no activity being indicated by 0 and severe activity by 10.
Change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score | Week 12
  The HAQ-DI assesses physical function in RA. The HAQ-DI score is the average of the highest score in each of eight categories. The total score is between 0-3.0, in 0.125 increments. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (218):
- United States (85):
  - AZ Arthritis and Rheumotology Research, PLLC - Flagstaff /ID# 253431, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Research - Glendale Office /ID# 255018, Glendale, Arizona
  - Sun Valley Arthritis Center Ltd. /ID# 254654, Peoria, Arizona
  - Arizona Arthritis & Rheumatology Associates - East Bell Road /ID# 253432, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates - East Bell Road /ID# 255021, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates - Tucson /ID# 255017, Tucson, Arizona
  - Arthritis and Rheumatism Associates /ID# 254013, Jonesboro, Arkansas
  - Providence - St. Jude Medical Center /ID# 252690, Fullerton, California
  - Newport Huntington Medical Group /ID# 252687, Huntington Beach, California
  - Purushotham & Akther Kotha MD, Inc /ID# 252704, La Mesa, California
  - Valerius Medical Group & Research Center of Greater Long Beach, Inc /ID# 252692, Los Alamitos, California
  - Rheumatology Center of San Diego /ID# 255038, San Diego, California
  - Millennium Clinical Trials /ID# 252689, Thousand Oaks, California
  - The Lundquist Institute at Harbor-UCLA Medical Center /ID# 252691, Torrance, California
  - Comprehensive Rheumatology Center /ID# 252688, Woodland Hills, California
  - University of Colorado Hospital /ID# 254617, Aurora, Colorado
  - Denver Arthritis Clinic /ID# 254058, Denver, Colorado
  - Tekton Research - Fort Collins - East Harmony Road /ID# 255036, Fort Collins, Colorado
  - Arthritis and Rheumatic Disease Specialties /ID# 260583, Aventura, Florida
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 253733, Boca Raton, Florida
  - Bay Area Arthritis and Osteo /ID# 254046, Brandon, Florida
  - Believe Clinical Trial /ID# 262355, Coral Springs, Florida
  - International Medical Research /ID# 254651, Daytona Beach, Florida
  - Omega Research Debary, LLC /ID# 253735, DeBary, Florida
  - Neoclinical Research /ID# 254622, Hialeah, Florida
  - Gnp Research - Hollywood /ID# 273563, Hollywood, Florida
  - Life Clinical Trials /ID# 256061, Margate, Florida
  - Lakes Research, LLC /ID# 255023, Miami, Florida
  - HMD Research LLC /ID# 253732, Orlando, Florida
  - Millennium Research /ID# 253744, Ormond Beach, Florida
  - Vitalia Research /ID# 274213, Palm Beach Gardens, Florida
  - BayCare Medical Group /ID# 253799, St. Petersburg, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 254649, Tampa, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 255264, Tampa, Florida
  - University of South Florida- Neuroscience Institute /ID# 253745, Tampa, Florida
  - Baycare Medical Group - Tampa /ID# 255268, Tampa, Florida
  - Atlanta Research Center For Rheumatology - Marietta /ID# 254623, Marietta, Georgia
  - Next Innovative Clinical Research - Chicago /ID# 273453, Chicago, Illinois
  - Deerbrook Medical Associates /ID# 254008, Libertyville, Illinois
  - OrthoIllinois /ID# 254057, Rockford, Illinois
  - Greater Chicago Specialty Physicians /ID# 254000, Schaumburg, Illinois
  - Clinic Of Dr. Robert Hozman/Clinical Investigation Specialists, Inc /ID# 253999, Skokie, Illinois
  - Willow Rheumatology and Wellness, PLLC /ID# 254712, Willowbrook, Illinois
  - Qualmedica Research - Evansville /ID# 254005, Evansville, Indiana
  - Western KY Rheumatology /ID# 255026, Hopkinsville, Kentucky
  - Bluegrass Community Research /ID# 254653, Lexington, Kentucky
  - Ochsner Health Center - The Grove /ID# 254059, Baton Rouge, Louisiana
  - The Arthritis & Diabetes Clinic, Inc. /ID# 254014, Monroe, Louisiana
  - Rheumatology Associates PA - Portland /ID# 255014, Portland, Maine
  - Beth Israel Deaconess Medical Center - Rheumatology /ID# 255029, Boston, Massachusetts
  - AA Medical Research Center - Grand Blanc /ID# 254007, Grand Blanc, Michigan
  - Advanced Rheumatology, PC /ID# 256059, Okemos, Michigan
  - St. Paul Rheumatology, PA /ID# 255037, Eagan, Minnesota
  - Arthritis Associates /ID# 253992, Hattiesburg, Mississippi
  - Kansas City Physician Partners /ID# 255035, Kansas City, Missouri
  - Clinvest Research LLC /ID# 254054, Springfield, Missouri
  - Logan Health Research - Glacier View Research Institute - Rheumatology /ID# 253738, Kalispell, Montana
  - Physician Research Collaboration, LLC /ID# 254012, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 253798, Lebanon, New Hampshire
  - Arthritis Rheumatic and Back Disease Associates. P.A. /ID# 255266, Voorhees Township, New Jersey
  - Arthritis and Osteoporosis Associates of New Mexico /ID# 252684, Las Cruces, New Mexico
  - NYU Langone Ambulatory Care Brooklyn Heights /ID# 254621, Brooklyn, New York
  - Joint And Muscle Research Institute /ID# 275128, Charlotte, North Carolina
  - Trinity Health Med Arts Clinic /ID# 254010, Minot, North Dakota
  - Paramount Medical Research and Consulting /ID# 254048, Middleburg Heights, Ohio
  - Rheumatology Associates of Oklahoma /ID# 253994, Oklahoma City, Oklahoma
  - Clinical Research of Philadelphia, LLC /ID# 255025, Philadelphia, Pennsylvania
  - West Tennessee Research Institute /ID# 254620, Jackson, Tennessee
  - Arthritis and Rheumatology Research Institute, PLLC /ID# 254045, Allen, Texas
  - Tekton Research, L.L.C /ID# 254004, Austin, Texas
  - Trinity Universal Research Associates - Carrollton /ID# 254648, Carrollton, Texas
  - Adriana Pop-Moody MD Clinic PA /ID# 255030, Corpus Christi, Texas
  - JPS Rheumatology Clinic /ID# 254050, Fort Worth, Texas
  - Biopharma Informatic - Houston - Business Center Drive /ID# 254051, Houston, Texas
  - Accurate Clinical Research - Houston /ID# 254647, Houston, Texas
  - Research Physicians Network, LLC /ID# 254053, Houston, Texas
  - R & H Clinical Research - 777 Katy /ID# 255024, Katy, Texas
  - West Texas Clinical Research /ID# 253736, Lubbock, Texas
  - Trinity Universal Research Associates, Inc /ID# 253995, Plano, Texas
  - Sun Research Institute /ID# 255019, San Antonio, Texas
  - Advanced Rheumatology of Houston /ID# 254003, The Woodlands, Texas
  - DM Clinical Research - Tomball /ID# 254001, Tomball, Texas
  - Rheumatology Clinic of Houston /ID# 254002, Tomball, Texas
  - Aurora Rheumatology and Immunotherapy Center /ID# 254049, Franklin, Wisconsin
  - Rheumatic Disease Center, LLP /ID# 254015, Glendale, Wisconsin
- Argentina (5):
  - Organizacion Medica de Investigacion (OMI) /ID# 253253, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Consultorios Reumatologicos Pampa /ID# 254095, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Aprillus Asistencia e Investigacion /ID# 253258, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Centro de Investigaciones Medicas Tucuman /ID# 253297, San Miguel de Tucumán, Tucumán Province
  - CIMER Centro Integral de Medicina Respiratoria /ID# 255277, San Miguel de Tucumán, Tucumán Province
- Belgium (4):
  - ReumaClinic /ID# 252277, Genk, Limburg
  - UZ Gent /ID# 252306, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan Brugge /ID# 252278, Bruges, West-Vlaanderen
  - Duplicate_CHU de Liege /ID# 252309, Liège
- Brazil (6):
  - CMiP - Centro Mineiro de Pesquisa Ltda - ME /ID# 254203, Juiz de Fora, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras /ID# 254201, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 254916, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 254202, Porto Alegre, Rio Grande do Sul
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 254917, São José do Rio Preto, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica /ID# 254200, São Paulo
- Bulgaria (7):
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 252354, Sofiya, Sofia
  - Diagnostic Consultative Centre (Dcc) - Foкus 5 /ID# 252555, Sofiya, Sofia
  - Umbal Kaspela /ID# 252343, Plovdiv
  - Medical center Unimed /ID# 252344, Plovdiv
  - MHAT Plovdiv /ID# 252342, Plovdiv
  - Diagnostic consultative center 17 Sofia /ID# 252341, Sofia
  - Military Medical Academy Multiprofile Hospital /ID# 252355, Sofia
- Canada (5):
  - Manitoba Clinic /ID# 254019, Winnipeg, Manitoba
  - Centre Rhumatologie de l'Est /ID# 254932, Rimouski, Quebec
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 253409, Sainte-Foy, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 256273, Trois-Rivières, Quebec
  - Dr. Latha Naik Medical Professional Corporation /ID# 254018, Saskatoon, Saskatchewan
- Chile (4):
  - Corporacion de Beneficiencia Osorno /ID# 252556, Osorno, Los Lagos Region
  - Centro Internacional de Estudios Clinicos - CIEC /ID# 252561, Santiago, Region Metropolitana Santiago
  - Clinica Dermacross /ID# 252560, Vitacura, Region Metropolitana Santiago
  - Complejo Asistencial Dr. Sotero del Rio /ID# 252559, Santiago, Santiago Metropolitan
- China (8):
  - The first affiliated hospital of bengbu medical college /ID# 252612, Bengbu, Anhui
  - Peking University First Hospital /ID# 252392, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 252393, Beijing, Beijing Municipality
  - The Third Affiliated Hospital, Sun Yat-Sen University /ID# 252394, Guangzhou, Guangdong
  - Zhuzhou Central Hospital /ID# 252390, Zhuzhou, Hunan
  - Nanjing Drum Tower Hospital /ID# 252613, Nanjing, Jiangsu
  - Jiangxi Pingxiang Peoples Hospital /ID# 252381, Pingxiang, Jiangxi
  - West China Hospital, Sichuan University /ID# 252364, Chengdu, Sichuan
- Colombia (5):
  - Hospital Pablo Tobón Uribe /ID# 253371, Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe SAS - Circaribe SAS /ID# 252587, Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y especialidades Medicas S.A.S- CIREEM /ID# 252586, Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S /ID# 252585, Zipaquirá, Cundinamarca
  - Fundacion Oftalmologica de Santander - FOSCAL /ID# 252589, Bucaramanga, Santander Department
- Croatia (5):
  - Medical Center Kuna-Peric /ID# 252452, Zagreb, City of Zagreb
  - Poliklinika Bonifarm /ID# 252741, Zagreb, City of Zagreb
  - Poliklinika Repromed /ID# 252451, Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 252453, Zagreb, City of Zagreb
  - Duplicate_Specijalna bolnica za medicinsku rehabilitaciju Krapinske Toplice /ID# 252455, Krapinske Toplice
- France (6):
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur /ID# 254224, Nice, Alpes-Maritimes
  - CHU Toulouse - Hopital Purpan /ID# 252402, Toulouse, Haute-Garonne
  - CHU Montpellier - Hôpital Lapeyronie /ID# 252386, Montpellier, Herault
  - CHU Amiens-Picardie Site Sud /ID# 252384, Amiens, Somme
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 252385, Orléans
  - Hôpital Charles-Nicolle /ID# 252908, Rouen
- Germany (5):
  - Rheumatologische-Immunologische Praxis Templin /ID# 252863, Templin, Brandenburg
  - Rheumazentrum Ruhrgebiet /ID# 252670, Herne, North Rhine-Westphalia
  - MVZ Rheumatologie und Autoimmunmedizin Hamburg GmbH /ID# 252667, Hamburg
  - Klinische Forschung im med. Versorgungsalltag GbR /ID# 254221, Planegg
  - Rheumazentrum Ratingen /ID# 252669, Ratingen
- Greece (3):
  - General Hospital of Athens Laiko /ID# 252258, Athens, Attica
  - University General Hospital Attikon /ID# 254751, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 252261, Heraklion, Crete
- Hungary (4):
  - Vital-Medicina Kft. /ID# 252399, Veszprém, Fejér
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 253311, Budapest
  - CMED Rehabilitacios es Diagnosztikai Kozpont /ID# 252400, Székesfehérvár
  - MÁV Kórház /ID# 252628, Szolnok
- Italy (3):
  - Azienda Ospedaliero Universitaria Careggi /ID# 252460, Florence, Firenze
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO /ID# 252461, Milan, Milano
  - Azienda Ospedaliero Universitaria delle Marche /ID# 252459, Ancona
- Japan (21):
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital /ID# 252836, Nagoya, Aichi-ken
  - Daido Clinic - Nagoya /ID# 253058, Nagoya, Aichi-ken
  - Kashiwa Kousei General Hospital /ID# 270033, Kashiwa-shi, Chiba
  - Sugimoto Rheumatology and Internal Medicine Clinic /ID# 252774, Fukui-shi, Fukui
  - Hamanomachi Hospital /ID# 253168, Fukuoka, Fukuoka
  - Shono Rheumatism Clinic /ID# 252591, Fukuoka, Fukuoka
  - Katayama Orthopedic Rheumatology Clinic /ID# 252746, Asahikawa-shi, Hokkaido
  - Sagawa Akira Rheumatology Clin /ID# 252773, Sapporo, Hokkaido
  - Hokkaido Medical Center For Rheumatic Diseases /ID# 270019, Sapporo, Hokkaido
  - Matsubara Mayflower Hospital /ID# 252834, Kato-shi, Hyōgo
  - Sanuki Municipal Hospital /ID# 252747, Sanuki-shi, Kagawa-ken
  - Bay Side Misato Medical Center /ID# 252661, Kochi, Kochi
  - Kumamoto Orthopaedic Hospital /ID# 253167, Kumamoto, Kumamoto
  - Medical Corporation Keiai Kai Clinic /ID# 252750, Miyazaki, Miyazaki
  - Sasebo Chuo Hospital /ID# 252662, Sasebo-shi, Nagasaki
  - Rinku Hashimoto Rheumatology Orthopaedics /ID# 270396, Izumisano, Osaka
  - St. Lukes International Hospital /ID# 253131, Chuo-ku, Tokyo
  - Keio University Hospital /ID# 253205, Shinjuku-ku, Tokyo
  - Tokito Clinic Rheumatology and Orthopaedics Surgery /ID# 253057, Shimonoseki-shi, Yamaguchi
  - Maeshima Rheumatology Clinic /ID# 270448, Ōita
  - Toyama Prefectural Central Hospital /ID# 270871, Toyama
- Mexico (5):
  - Centro Integral en Reumatologia S.A de C.V /ID# 252872, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 253480, Guadalajara, Jalisco
  - Hospital de Jesus /ID# 253114, Mexico City, Mexico City
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 252873, Mexico City, Mexico City
  - Investigacion y Biomedicina de Chihuahua /ID# 253115, Chihuahua City
- Portugal (3):
  - Hospital Garcia de Orta /ID# 252491, Almada, Setúbal District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 252489, Ponte de Lima, Viana do Castelo District
  - Unidade Local de Saude de Santa Maria, EPE /ID# 252492, Lisbon
- Puerto Rico (2):
  - GCM Medical Group PSC /ID# 252700, San Juan
  - Mindful Medical Research /ID# 252693, San Juan
- Romania (5):
  - Cabinet Medical Dr. Avram S.R.L /ID# 254133, Timișoara, Timiș County
  - Banat Carina Med SRL /ID# 252757, Timișoara, Timiș County
  - Spitalul Judetean de Urgenta Bacau /ID# 252860, Bacau
  - Spitalul Clinic Sf. Maria /ID# 252759, Bucharest
  - Spitalul Clinic Sf. Maria /ID# 253334, Bucharest
- Serbia (6):
  - Institute for Rheumatology /ID# 252333, Belgrade, Beograd
  - Institute for Rheumatology /ID# 252334, Belgrade, Beograd
  - Institute for Rheumatology /ID# 252335, Belgrade, Beograd
  - Institute for Rheumatology /ID# 252338, Belgrade, Beograd
  - Special Hospital for Rheuma /ID# 252336, Novi Sad, Vojvodina
  - Special Hospital for Rheuma /ID# 252339, Novi Sad, Vojvodina
- South Africa (7):
  - University of Pretoria /ID# 252368, Pretoria, Gauteng
  - Dr Elsa van Duuren /ID# 252387, Pretoria, Gauteng
  - Emmed Research cc /ID# 254317, Pretoria, Gauteng
  - Dr Asokan Naidoo /ID# 252894, Umhlanga, KwaZulu-Natal
  - Winelands Medical Research - Somerset West /ID# 252745, Cape Town, Western Cape
  - Arthritis Clinical Research Trials /ID# 252370, Cape Town, Western Cape
  - Winelands Medical Research Centre /ID# 252369, Stellenbosch, Western Cape
- South Korea (5):
  - SoonChunHyang University Hospital Cheonan /ID# 254942, Cheonan-si, Chungcheongnam-do
  - Chungnam National University Hospital /ID# 252159, Daejeon, Daejeon Gwang Yeogsi
  - Chonnam National University Bitgoeul Hospital /ID# 254802, Gwangju, Gwangju Gwang Yeogsi
  - Seoul National University Hospital /ID# 252160, Seoul, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospital /ID# 252161, Seoul, Seoul Teugbyeolsi
- Spain (5):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 252430, Santiago de Compostela, A Coruna
  - Hospital Marina Baixa /ID# 254141, Villajoyosa, Alicante
  - Hospital Universitario Germans Trias i Pujol /ID# 254144, Badalona, Barcelona
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 252425, Sabadell, Barcelona
  - Hospital Universitario y Politecnico La Fe /ID# 254143, Valencia
- United Kingdom (4):
  - Royal Free Hospital /ID# 252297, London, Greater London
  - The Queen Elizabeth Hospital, Kings Lynn NHS Foundation Trust /ID# 252301, Kings Lynn, Norfolk
  - Queen Mary University of London /ID# 252671, London
  - Portsmouth Hospitals University NHS Trust /ID# 252772, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-700